CLINICAL TRIAL: NCT06999408
Title: A Prospective, 8-Month, Randomized Pilot Study of TargetCool™ Cryo-Modulation and BENEV Exosome Regenerative Complex+® for Hair Density Enhancement in Adults With Non-Scarring Hair Thinning
Brief Title: Efficacy and Safety of TargetCool + Benev Exosomes in Patients With Hair Thinning
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Recens Medical, Inc. (Industry)
Collaborators: Benev Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-2025-DERM-001-IIT
Record Dates: First submitted 2025-05-14; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hair Diseases; Alopecia; Hair Thinning
Keywords: Exosomes; TargetCool; Hair thinning; mirconeedling
MeSH Terms: conditions — Hair Diseases; Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- TargetCool with Benev exosome Boost (Active Comparator)
  Interventions: Device: Scalp tattoo; Device: Canfield HairMetrix®; Device: TargetCool
- Microneedling followed by TargetCool Boosting with Benev exosome (Active Comparator)
  Interventions: Device: Scalp tattoo; Device: Canfield HairMetrix®; Device: TargetCool; Device: Microneedle-facilitated lidocaine application
- Microneedling to depth of 0.5mm followed by Benev exosome topical (Active Comparator)
  Interventions: Device: Scalp tattoo; Device: Canfield HairMetrix®; Device: Microneedle-facilitated lidocaine application

INTERVENTIONS:
Device: Scalp tattoo — A micropigmentation scalp tattoo will be applied at baseline to mark consistent photographic sites.
Device: Canfield HairMetrix® — Canfield HairMetrix® imaging will be utilized to capture global and trichoscopic hair measurements.
Device: TargetCool — Boosting will be used to apply exosomes
  Arms: Microneedling followed by TargetCool Boosting with Benev exosome; TargetCool with Benev exosome Boost
Device: Microneedle-facilitated lidocaine application — Microneedling will be performed to a depth of 0.5 mm.
  Arms: Microneedling followed by TargetCool Boosting with Benev exosome; Microneedling to depth of 0.5mm followed by Benev exosome topical

SUMMARY:
This clinical trial is testing a new approach to help improve hair thinning using a combination of cosmetic treatments. The purpose of the study is to learn whether applying exosomes to the scalp, along with microneedling and a precision cooling device called TargetCool™. This study aims to determine whether this combination approach offers synergistic benefits for individuals with hair thinning.

Exosomes are tiny particles that come from stem cells and contain growth factors and other nutrients. They are being studied for their potential to help regenerate skin and hair. TargetCool™ is an FDA-cleared device that uses precision cooling to reduce inflammation and improve comfort. Microneedling is a common, minimally invasive procedure that uses small needles to stimulate the skin and help absorb topical products more effectively.

The study will include healthy men (ages 18 to 70) and women (ages approximately 45 to 70) who are not of childbearing potential. A total of 9 to 15 participants will be randomly placed into one of three groups:

Group 1: Exosomes with TargetCool™ Group 2: Microneedling followed by exosomes and TargetCool™ Group 3: Microneedling followed by exosomes only Participants will receive four treatments over 9 weeks. Each visit may include microneedling, TargetCool™ treatment, and exosome application depending on group assignment. A small tattoo will be placed on the scalp to help capture consistent photographs, and a special imaging system (Canfield HairMetrix®) will be used to measure hair changes.

Participants will return for follow-up visits at 3 and 6 months after the final treatment. The results will help determine whether this combination of cosmetic treatments is safe and beneficial for people experiencing hair thinning.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males between 18-70 years of age and females not of child-bearing age 45-70 years of age of all Fitzpatrick Skin Types.
2. Subjects must be willing to provide verbal understanding and sign an Informed Consent Form, HIPAA Form and Photography Release Form approved by the Institutional Review Board.
3. Subjects must be in general good health, as determined by the Investigator.
4. Subjects with hair thinning as determined on initial study assessment by the Investigator.
5. Patients are not on medical treatment or have been on stable treatment for >12 months (eg. minoxidil, finasteride, dutasteride, PRP, LLLT)
6. Subjects willing to not substantially change their current diet, medications, or exercise routines for the duration of the study. If a subject receives physician guidance during the study to change diet, medications, or exercise routine, the subject will need to notify the clinic as soon as possible.
7. Subjects willing to have Canfield digital photography of the entire head/hair region for overall evaluation of general hair growth and quality by the Investigator.
8. Subjects willing to have TargetCool boosting or microneedling of the scalp region with or followers by application of exosomes.
9. Subjects must be willing and able to complete and understand the rating questionnaires.
10. Subjects must be willing and able to attend all study visits and comply with the post procedure and lifestyle instructions

Exclusion Criteria:

1. Subjects who are of child-bearing age, pregnant, nursing mothers, planning a pregnancy during the course of the study, or become pregnant during the study.
2. Subjects who have had a hair transplant.
3. Subjects who have recently (within the last 3 months) started the use of hormones for birth control or hormone replacement therapy (HRT). Women currently using hormones for birth control or HRT must have been on a stable dose (3 months or longer) in order to be eligible for the study.
4. Subjects who started any new hair loss treatment in the last 12 months.
5. Subjects who have used prescription drugs known to affect the hair growth cycle within the last 3 months (e.g., hormone-based birth control for less than 12 months, cyproterone acetate, aldactone/spironolactone or any 5-alpha-reductase inhibitor).
6. Subjects who have regularly used anti-androgenic therapies (i.e. spironolactone, flutamide, cyproterone acetate, progesterone and/or bicalutamide) or undergone any other hair or scalp treatments within the last 12 months.
7. Subjects suffering from other hair loss disorders, such as alopecia areata, scarring alopecia, and telogen effluvium as determined during initial study assessment and physical exam by the Investigator.
8. Subjects with self-reported uncontrolled diseases (i.e. diabetes, hypertension, hyperthyroidism, hypothyroidism, etc.). Whether medical conditions are under control with or without treatment will be assessed on an individual basis by the Investigator based on her medical and clinical expertise.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Terminal Hair Counts | 32 weeks (8 months)
  Terminal hair is defined as coarse hair, short or long, found on the scalp with minimum cross-sectional diameter of 40 micrometers. This is calculated by the Canfield HairMetrix System.
Change in Vellus Hair Counts | 32 weeks (8 months)
  Vellus hair is defined as fine, short hairs found on the scalp with maximum cross-sectional diameter of 40 micrometers. This is calculated by the Canfield HairMetrix System.
Change in Total Hair Counts | 32 weeks (8 months)
  Total hairs equals the sum of Terminal and Vellus hairs in the target area. This is calculated by the Canfield HairMetrix System.
Change in average hair width | 32 weeks (8 months)
  This is the average hair width calculated in micrometers by the Canfield HairMetrix System.

SECONDARY OUTCOMES:
Change in Investigator Hair Growth Global Improvement Scale | 32 weeks (8 months)
  The treating Investigator will complete this assessment by circling the number on the scale that corresponds to the description that best fits the current global growth improvement at delineated visits as indicated in the schedule of events, compared to baseline. The Investigator will complete this assessment at the end of study. The Investigator must complete this assessment using global photographs obtained compared to baseline. In addition, the Investigator may use their clinical judgment from the in-person visit.
  3 Greatly worsened 2 Moderately worsened
  1 Slightly worsened 0 No change
  1. Slightly improved
  2. Moderately improved
  3. Greatly improved
Change in Subject Hair Self-Assessment Questionnaire scores | 32 weeks (8 months)
  Overall hair appearance:
  1. Greatly Decreased/Worsened
  2. Moderately Decreased/Worsened
  3. Slightly Decreased/Worsened
  4. No Change
  5. Slightly Increased/Improved
  6. Moderately Increased/ Improved
  7. Greatly Increased/ Improved
Change in Hair Treatment Subject Satisfaction Questionnaire scores | 32 weeks (8 months)
  1. How satisfied are you with this treatment for your thinning hair? 5 = Very Satisfied 4 = Satisfied 3 = Neutral 2 = Dissatisfied 1 = Very Dissatisfied
  2. How satisfied are you with the overall health of your hair after this treatment? 5 = Very Satisfied 4 = Satisfied 3 = Neutral 2 = Dissatisfied 1 = Very Dissatisfied
  3. Overall, how satisfied are you with the ease of this treatment? 5 = Very Satisfied 4 = Satisfied 3 = Neutral 2 = Dissatisfied 1 = Very Dissatisfied
  4. Overall, now that you have tried this treatment and completed the study, how likely are you to continue the treatment in the future? 5 = Very Likely 4 = Somewhat Likely 3 = Neutral 2 = Somewhat Unlikely 1 = Very Unlikely
  5. Overall, how likely are you to recommend this treatment to a family member or friend? 5 = Very Likely 4 = Somewhat Likely 3 = Neutral 2 = Somewhat Unlikely 1 = Very Unlikely

OTHER OUTCOMES:
Frequency of both local and systemic Adverse Events | 32 weeks (8 months)
  An adverse event is any adverse change from the subject's baseline condition, i.e. any subjective signs and symptoms, or change in a concomitant disease present at the screening visit. This includes inter-current signs, symptoms, illness and significant deviations from baseline which may occur during the course of the clinical study, whether considered related to treatment or not.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Avram, MD, Principal Investigator; Dawn Queen, MD, Principal Investigator
Locations (1):
- Marc Avram MD, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this study will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 6 months after publication and available for up to 2 years.
Access Criteria: Requests must include a brief proposal outlining study aims and methodology. The study team will review each request for scientific merit. Data will be shared via secure, password-protected transfer.
  Researchers may request access by contacting michele@dravram.com.

REFERENCES:
- [Background] Ha DH, Kim SD, Lee J, Kwon HH, Park GH, Yang SH, Jung JY, Lee JH, Park SR, Youn J, Lee SH, Kim JE, Lim J, Lee HK, Cho BS, Yi YW. Toxicological evaluation of exosomes derived from human adipose tissue-derived mesenchymal stem/stromal cells. Regul Toxicol Pharmacol. 2020 Aug;115:104686. doi: 10.1016/j.yrtph.2020.104686. Epub 2020 May 22. PMID 32450131
- [Background] Ersan M, Ozer E, Akin O, Tasli PN, Sahin F. Effectiveness of Exosome Treatment in Androgenetic Alopecia: Outcomes of a Prospective Study. Aesthetic Plast Surg. 2024 Nov;48(21):4262-4271. doi: 10.1007/s00266-024-04332-3. Epub 2024 Aug 22. PMID 39174804
- [Background] Zhou Y, Seo J, Tu S, Nanmo A, Kageyama T, Fukuda J. Exosomes for hair growth and regeneration. J Biosci Bioeng. 2024 Jan;137(1):1-8. doi: 10.1016/j.jbiosc.2023.11.001. Epub 2023 Nov 23. PMID 37996318
- [Background] Kost Y, Muskat A, Mhaimeed N, Nazarian RS, Kobets K. Exosome therapy in hair regeneration: A literature review of the evidence, challenges, and future opportunities. J Cosmet Dermatol. 2022 Aug;21(8):3226-3231. doi: 10.1111/jocd.15008. Epub 2022 Jun 2. PMID 35441799
- [Background] Gupta AK, Wang T, Rapaport JA. Systematic review of exosome treatment in hair restoration: Preliminary evidence, safety, and future directions. J Cosmet Dermatol. 2023 Sep;22(9):2424-2433. doi: 10.1111/jocd.15869. Epub 2023 Jun 28. PMID 37381168
- [Background] Queen D, Avram MR. Exosomes for Treating Hair Loss: A Review of Clinical Studies. Dermatol Surg. 2025 Apr 1;51(4):409-415. doi: 10.1097/DSS.0000000000004480. Epub 2024 Oct 24. PMID 39447204
- See also: TargetCool — https://coolhealth.com
- See also: Exosome Regenerative Complex+ — https://benev.com